CLINICAL TRIAL: NCT06658990
Title: Effect of Ultrasound Positioning Assisted Cheek Needle Therapy on Postoperative Recovery Quality of Patients with Radical Resection of Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024ky042
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-08

CONDITIONS: Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- buccal acupuncture (Experimental)
  Interventions: Procedure: buccal acupuncture
- control (Active Comparator)
  Interventions: Drug: control

INTERVENTIONS:
Procedure: buccal acupuncture — ultrasound positioning assisted buccal acupuncture
  Arms: buccal acupuncture
Drug: control — Sufentanil is used after surgery
  Arms: control

SUMMARY:
To explore the effect of ultrasound positioning assisted buccal acupuncture on postoperative pain and recovery quality of patients undergoing thoracoscopic radical resection

ELIGIBILITY:
Inclusion Criteria:

1. Tracheal intubation under general anesthesia
2. Young and middle-aged patients aged 18-65 years
3. BMI: 18.5-28kg /m2

Exclusion Criteria:

1. head and facial trauma, infection, disease
2. more than 2 kinds of coronary heart disease, hypertension, stroke, diabetes, immune disease and other diseases before surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Number of additional analgesics | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Wang Mengyao, Yangzhou, Jiangsu, China